CLINICAL TRIAL: NCT06763588
Title: Changes in Diet Quality After Bariatric Surgery Measured With the 'Eetscore' Screener.
Brief Title: Diet Quality Before and After Metabolic Bariatric Surgery (Eetscore Study)
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Wageningen University & Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-1214
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Overweight; Bariatric Surgery; Nutrition Assessment; Diet Quality
Keywords: Screener; Diet quality; Obesity; Metabolic bariatric surgery; Weight loss surgery; Validity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to learn more about the use of a short screener for diet quality (Eetscore FFQ) in bariatric patients and about changes in diet quality before and after the bariatric procedure.

ELIGIBILITY:
Inclusion Criteria:

* Approved for (primary) bariatric surgery
* Aged 18-65 years
* Following the standard care pathway

Exclusion Criteria:

* Previous bariatric procedure other than adjustable gastric banding
* Non-Dutch eating pattern
* Active eating disorders
* Inability to fill in questionnaires or food records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe obesity who were eligible and scheduled for metabolic bariatric surgery at Vitalys Obesity Clinic, part of Rijnstate hospital (Arnhem, the Netherlands), were asked to participate in this prospective cohort study. Participants were included approximately 6 weeks pre-surgery and followed up until 5 years post-surgery.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Dutch Healthy Diet index score | Before surgery and at 6 mo after surgery
  The DHD2015-index consists of fifteen components representing the Dutch food-based dietary guidelines of 2015: vegetables, fruit, wholegrain products, legumes, nuts, dairy, fish, tea, fats and oils, coffee, red meat, processed meat, sweetened beverages, alcohol and Na. Additionally, the component 'unhealthy food choices' was added based on the guideline of the Netherlands Nutrition Centre. For every component, the score ranges from 0 (no adherence) to 10 points (complete adherence), resulting in a total score between 0 and 160 points.
  Total DHD2015-index score and individual component scores were calculated from the Eetscore FFQ and 3-day food records.

SECONDARY OUTCOMES:
Macro- and micronutrient intake | Before surgery and at 6 mo after surgery
  Macronutrient composition of the diet was evaluated by intake of total energy, total carbohydrates and mono- and disaccharides, total protein, plant-based and animal-based protein, total fat, saturated fat, monounsaturated fatty acids and polyunsaturated fatty acids (including alpha-linolenic acid, eicosapentaenoic acid, and docosahexaenoic acid), and dietary fibre. Furthermore, dietary intake of a limited range of micronutrients for which bariatric patients often display low serum levels was assessed: folate, vitamin B12, vitamin D, calcium and iron.
Dietary intake at 3 and 5 years post-surgery | 3 y and 5 y after surgery
  Dutch Healthy Diet index score + micro- and macronutrient intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Vitalys/Rijnstate, Elst, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heusschen L, Berendsen AAM, Balvers MGJ, Deden LN, de Vries JHM, Hazebroek EJ. Changes in nutrient composition and diet quality in the first 6 months following bariatric surgery: An observational cohort study. J Hum Nutr Diet. 2024 Feb;37(1):365-376. doi: 10.1111/jhn.13258. Epub 2023 Nov 14. PMID 37964680
- [Result] Heusschen L, Berendsen AA, Balvers MG, Deden LN, de Vries JH, Hazebroek EJ. Relative validity of a short screener to assess diet quality in patients with severe obesity before and after bariatric surgery. Public Health Nutr. 2022 Jul 4;25(10):1-11. doi: 10.1017/S1368980022001501. Online ahead of print. PMID 35786490